CLINICAL TRIAL: NCT05850351
Title: The Effect of 12-Week-Virtual Reality Based Tele-Exercises on Exercise Capacity in Cystic Fibrosis Patients: A Randomized Controlled, Single (Assessor)-Blind Study
Brief Title: Virtual Reality Based Tele-Exercises on Exercise Capacity in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ozden Ozyemisci Taskiran, Clinical Professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.153.IRB1.056
Record Dates: First submitted 2023-04-17; First posted 2023-05-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis in Children; Telerehabilitation; Virtual Reality
Keywords: Cystic Fibrosis; Aerobic Exercise; Telerehabilitation; Virtual Reality
MeSH Terms: conditions — Cystic Fibrosis | interventions — Pharmaceutical Services, Online

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the study, outcomes assessor will not know which group the children belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Children with cystic fibrosis will be given exercise in the form of a game in a virtual environment in groups of 4-6 children, accompanied by a physiotherapist, for 12 weeks, 3 days a week, between 30-45 minutes.
  Interventions: Other: Virtual reality
- Online (Experimental): Children with cystic fibrosis will be given online aerobic exercise for 12 weeks, 3 days a week, 30-45 minutes, in groups of 4-6 children, accompanied by a physiotherapist.
  Interventions: Other: Online

INTERVENTIONS:
Other: Virtual reality — Virtual reality is a simulated experience that creates a virtual environment to give the user the feeling of an immersive virtual world, using glasses and a handheld device that can track hand movements. Activities that will improve the functional and respiratory capacity of children with cystic fibrosis will be developed and integrated into the virtual reality game.
  Arms: Virtual reality
Other: Online — Online exercises are physical activities that are performed via a video-conferencing tool. Children will be at their home environment and exercises which will improve their functional and respiratory capacity will be instructed and supervised by a physiotherapist.
  Arms: Online

SUMMARY:
The goal of this clinical trial is to investigate the effects of a-12-week virtual reality exercise program, applied as tele-exercise, on the exercise capacity of children with cystic fibrosis, whose physical activity level is further restricted during the pandemic. The main questions it aims to answer are:

Does aerobic tele-exercise increase functional capacity in cystic fibrosis patients? Will there be a difference in treatment outcomes between the virtual reality group and the online exercise group?

Participants will be randomized into two groups; virtual reality group and online group. Physical activity will be provided to the virtual reality group in the form of team activities in a virtual environment, and the other group will be provided online exercises at their home. For this purpose, virtual reality headsets will be provided to patients to give the impression of a natural, immersive environment and realistic experience.

Researchers will compare exercise compliance and functional capacity between the virtual reality group and the online group.

DETAILED DESCRIPTION:
This project aims to investigate the effects of a-12-week virtual reality exercise program, applied as tele-exercise, on the exercise capacity of children with cystic fibrosis, whose physical activity level is further restricted during the pandemic. The originality of this study is that it would be the first study in which immersive virtual reality exercises will be performed through tele-exercise in cystic fibrosis.

Prognosis in cystic fibrosis is related to respiratory capacity and physical activity level. Aerobic exercise positively affects lung functions; increases aerobic capacity, survival and quality of life in cystic fibrosis.

Face-to-face activities in children with cystic fibrosis increase the risk of cross-contamination and lung infection. Remote exercises will be more cost effective in terms of transportation/time loss as well as reduction of infection risk.

Virtual reality exercises based on video game activities provide a good alternative, especially for motivating and increasing the adaptation of young individuals to rehabilitation. This project plans to investigate the hypothesis that exercise capacities would increase with virtual reality exercises performed in groups that help socialization, without the risk of hospital infection.

Patients will be randomized into two groups. Physical activity will be provided to the virtual reality group in the form of team activities in a virtual environment. For this purpose, virtual reality headsets will be provided to patients to give the impression of a natural, immersive environment and realistic experience. The activities will be carried out in groups of 4-6 children with cystic fibrosis, accompanied by a physiotherapist, for 12 weeks, 3 days a week, between 30-45 minutes in both groups.

At the beginning and end of the 12-week program, patients will be evaluated. The 6-minute walk test will be used to measure exercise capacity in children with cystic fibrosis. At the end of the treatment, it is expected that children with cystic fibrosis in the virtual reality group will reach as high exercise capacity as the other group.

ELIGIBILITY:
Inclusion Criteria:

* 12 and 16 years,
* Clinical stability without disease exacerbations in the 4 weeks prior to their enrollment into the study
* Having access to internet and parental or legal caregiver consent

Exclusion Criteria:

* Children with a pulmonary exacerbation in the previous 4 weeks,
* Active pulmonary infection,
* Evidence of pulmonary hypertension
* Any cardiological, musculoskeletal, neurological or cognitive comorbidities that prevent exercise participation,
* Behavioral ot intellectual difficulties that prevent participation in assessments or exercises provided remotely
* Children with oxygen supplementation (daily continuous use or > 2 L/min at night)
* Lung transplant candidates

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance | 12 weeks
  6-minute walk distance is a valid and reproducible test in the assessment of functional capacity in children and adolescent with cystic fibrosis. The children were asked to walk in a 30-meter corridor as far as possible in 6 minutes. Distance covered in 6 minutes was recorded as the primary outcome measure.

SECONDARY OUTCOMES:
Hand grip strength | 12 weeks
  Hand grip strength is an indicator of overall muscle strength and will be measured using a dynamometer. Maximum of the six trials and the dominance of hand with the maximum measurement will be recorded in kg.
Quadriceps strength | 12 weeks
  Quadriceps strength will be measured using the digital dynamometer. Strength will be measured in both limbs.
Deltoid strength | 12 weeks
  Deltoid strength will be measured using the digital dynamometer. Strength will be measured in both limbs.
Cystic Fibrosis Questionnaire-Revised | 12 weeks
  Health-related quality of life was assessed using Cystic Fibrosis Questionnaire-Revised. Items are scored using a 4-point Likert scale. Total score ranges between 0 to 100. Higher scores indicate better quality of life. The questionnaire operates under 9 quality of health domains (physical functioning, role functioning, vitality, emotional functioning, social functioning, body image, eating problems, treatment burden and school functioning), 1 health perception (health perception) and 3 symptom domains (weight, respiratory and digestive symptoms).
Forced expiratory volume | 12 weeks
  Pulmonary function test will be assessed using a spirometry according to the guideline of American Thoracic Society. Forced expiratory volume in 1 second will be recorded.
Forced vital capacity | 12 weeks
  Pulmonary function test will be assessed using a spirometry according to the guideline of American Thoracic Society. Forced vital capacity will be recorded
Forced expiratory volume/Forced vital capacity | 12 weeks
  Pulmonary function test will be assessed using a spirometry according to the guideline of American Thoracic Society. Forced expiratory volume/Forced vital capacity will be recorded
The Physical Activity Questionnaire | 12 weeks
  To assess the level of physical activity in children, The Physical Activity Questionnaire for Older Children and adolescents will be used, which consist of 10 and 9 items, respectively. First item asks frequency of participation in 14 and 22 common leisure and sport activities in the past 7 days, respectively. Each item is scored on a 5-point rating scale and a mean score for the first item is calculated. Total score is the mean of scores of all items (1: low level of physical activity and 5: high level of physical activity)
System Usability Scale | up to 12 weeks
  To evaluate the virtual reality or online exercise experience Turkish translation of the System Usability Scale will be applied.
The Physical Activity Enjoyment Scale | up to 12 weeks
  The Physical Activity Enjoyment Scale- short scale consists of 8 items. It will be used to assess the pleasure from physical activity. Each item is scored rated on a 7-point Likert-type scale (1: strongly disagree to 7: strongly agree).
Accelerometer | 12 weeks
  All participants will be asked to wear Actiwatch-2 wrist accelerometer to measure activity.
  It records and stores the time and the intensity of movements. Actiwatch data will be transferred offline to a computer and automatically stored in activity counts by date and time using a software. Participants will wear the actiwatch continuously on the wrist of their non-dominant hand, removing the device only for activities involving water..
Body weight | 12 weeks
  Body weight will be measured as kilograms with Bioimpedance analysis.
Body height | 12 weeks
  Body height will be measured as meters with Bioimpedance analysis.
Body mass index | 12 weeks
  Body mass index z score will be calculated by adjusting weight and height values measured according to age and gender of the children as kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Prof
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade Lima C, Dornelas de Andrade A, Campos SL, Brandao DC, Mourato IP, Britto MCA. Six-minute walk test as a determinant of the functional capacity of children and adolescents with cystic fibrosis: A systematic review. Respir Med. 2018 Apr;137:83-88. doi: 10.1016/j.rmed.2018.02.016. Epub 2018 Feb 26. PMID 29605218
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Bhatia R, Kaye M, Roberti-Miller A. Longitudinal assessment of exercise capacity and quality of life outcome measures in cystic fibrosis: A year-long prospective pilot study. J Eval Clin Pract. 2020 Feb;26(1):236-241. doi: 10.1111/jep.13105. Epub 2019 Feb 13. PMID 30761692
- [Background] Hommerding PX, Donadio MV, Paim TF, Marostica PJ. The Borg scale is accurate in children and adolescents older than 9 years with cystic fibrosis. Respir Care. 2010 Jun;55(6):729-33. PMID 20507656
- [Background] Bellini SG, Chapman P, Szendre K, McDonald C, Williams N, Hopkin L, Eggett D, Dean A. Changes in handgrip strength in children with cystic fibrosis compared to children without cystic fibrosis. Clin Nutr ESPEN. 2021 Apr;42:206-211. doi: 10.1016/j.clnesp.2021.01.038. Epub 2021 Feb 9. PMID 33745579
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Bohannon RW, Wang YC, Bubela D, Gershon RC. Handgrip Strength: A Population-Based Study of Norms and Age Trajectories for 3- to 17-Year-Olds. Pediatr Phys Ther. 2017 Apr;29(2):118-123. doi: 10.1097/PEP.0000000000000366. PMID 28350764
- [Background] Bobos P, Nazari G, Lu Z, MacDermid JC. Measurement Properties of the Hand Grip Strength Assessment: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2020 Mar;101(3):553-565. doi: 10.1016/j.apmr.2019.10.183. Epub 2019 Nov 13. PMID 31730754
- [Background] Villafane JH, Valdes K, Bertozzi L, Negrini S. Minimal Clinically Important Difference of Grip and Pinch Strength in Women With Thumb Carpometacarpal Osteoarthritis When Compared to Healthy Subjects. Rehabil Nurs. 2017 May/Jun;42(3):139-145. doi: 10.1002/rnj.196. PMID 25557054
- [Background] Sole A, Olveira C, Perez I, Hervas D, Valentine V, Baca Yepez AN, Olveira G, Quittner AL. Development and electronic validation of the revised Cystic Fibrosis Questionnaire (CFQ-R Teen/Adult): New tool for monitoring psychosocial health in CF. J Cyst Fibros. 2018 Sep;17(5):672-679. doi: 10.1016/j.jcf.2017.10.015. Epub 2017 Nov 20. PMID 29157922
- [Background] Quittner AL, Sawicki GS, McMullen A, Rasouliyan L, Pasta DJ, Yegin A, Konstan MW. Psychometric evaluation of the Cystic Fibrosis Questionnaire-Revised in a national sample. Qual Life Res. 2012 Sep;21(7):1267-78. doi: 10.1007/s11136-011-0036-z. Epub 2011 Oct 14. PMID 21993695
- [Background] Crocker PR, Bailey DA, Faulkner RA, Kowalski KC, McGrath R. Measuring general levels of physical activity: preliminary evidence for the Physical Activity Questionnaire for Older Children. Med Sci Sports Exerc. 1997 Oct;29(10):1344-9. doi: 10.1097/00005768-199710000-00011. PMID 9346166
- [Background] Erdim L, Ergun A, Kuguoglu S. Reliability and validity of the Turkish version of the Physical Activity Questionnaire for Older Children (PAQ-C). Turk J Med Sci. 2019 Feb 11;49(1):162-169. doi: 10.3906/sag-1806-212. PMID 30764593
- [Background] Mullen SP, Olson EA, Phillips SM, Szabo AN, Wojcicki TR, Mailey EL, Gothe NP, Fanning JT, Kramer AF, McAuley E. Measuring enjoyment of physical activity in older adults: invariance of the physical activity enjoyment scale (paces) across groups and time. Int J Behav Nutr Phys Act. 2011 Sep 27;8:103. doi: 10.1186/1479-5868-8-103. PMID 21951520
- [Derived] Ozyemisci Taskiran O, Albayrak H, Kog C, Atli E, Gonullu E, Yantac AE, Uyan ZS. The effect of a 12-week tele-exercise using immersive virtual reality on functional capacity in adolescents with cystic fibrosis: A randomized controlled, single (assessor) - blind study. Respir Med. 2025 Nov;248:108362. doi: 10.1016/j.rmed.2025.108362. Epub 2025 Sep 20. PMID 40983137